CLINICAL TRIAL: NCT04695197
Title: Malaria as a Risk Factor for COVID-19 in Western Kenya and Burkina Faso
Acronym: MALCOV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Kenya Medical Research Institute (Other); Groupe de Recherche Action en Sante (Other); Centres for Disease Control and Prevention, Kenya. (Other); Bill and Melinda Gates Foundation (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-063; 202009642148520 (Registry Identifier: Pan African Clinical Trial Registry (PACTR))
Record Dates: First submitted 2020-12-14; First posted 2021-01-05 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2021-02

CONDITIONS: Covid-19; Malaria
MeSH Terms: conditions — COVID-19; Malaria | interventions — Artemether, Lumefantrine Drug Combination; pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Intervention Model Description: Permuted block randomization
Masking Description: Masking: blinding of primary outcome assessor (off-site laboratory-based staff)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artemether-lumefantrine (Active Comparator): Artemether-lumefantrine, standard 3-day antimalarial treatment regimen.
  Interventions: Drug: Artemether-lumefantrine (AL)
- Pyronaridine-artesunate (Experimental): Pyronaridine-artesunate, standard 3-day antimalarial treatment regimen.
  Interventions: Drug: Pyronaridine-artesunate (PA)

INTERVENTIONS:
Drug: Artemether-lumefantrine (AL) — Current first line treatment of malaria. Dose: Bodyweight (kg) Dose (mg) of artemether + lumefantrine given twice daily for 3 days (total, six doses) 5 to < 15 20 + 120 15 to < 25 40 + 240 25 to < 35 60 + 360 >=35 80 + 480; Twice daily for 3 days (total, six doses)
  Other Names: Coartem
  Arms: Artemether-lumefantrine
Drug: Pyronaridine-artesunate (PA) — Antimalarial; Dose: Body weight (kg) Dose (mg) of pyronaridine + aresunate given once daily for 3 days (total, three doses) 5 to < 8 60 + 20 8 to <15 120 + 40 15 to <20 180 + 60 20 to <24 kg 180 + 60 24 to <45 360 + 120 45 to <65 540 + 180 >=65 720 + 240; Once-daily for 3 days (total, three doses).
  Other Names: Pyramax
  Arms: Pyronaridine-artesunate

SUMMARY:
It is unknown whether malaria or malaria treatment affects COVID-19 severity, immune responses to SARS-CoV-2 virus, or viral loads and/or duration of shedding and therewith the onwards spread of SARS-COV-2. An observational cohort study will be conducted in 708 newly diagnosed COVID-19 patient of all ages in western Kenya and Burkina-Faso. They will be enrolled in hospitals with COVID-19 testing facilities from a source population screened for SARS-CoV-2 (N~4,720). Approximately 142 of the 708 COVID-19 patients are expected to be co-infected with malaria. They will be enrolled in the nested malaria treatment trial and randomized to receive 3-days of artemether-lumefantrine (the current standard of care) or pyronaridine-artesunate, a highly effective antimalarial with known antiviral properties against SARS-CoV-2 in-vitro, that is newly registered and being rolled out in Africa. Disease progression will be assessed and nasal swabs and blood samples will be taken during home/clinic visits on days 1, 3, 7, 14, 21, 28, and 42. Patients self-isolating will be phoned daily in between scheduled visits for the first 14 days to assess signs and symptoms. Hospitalisation, self-isolation and home-based care will follow national guidelines. The WHO clinical progression scale and FLU-PRO plus scales will be used to compare disease progression between COVID-19 patients with and without malaria, and by malaria. Other endpoints include seroconversion/reversion rates, chemokine/cytokine responses, T and B cell responses, viral load and duration of viral carriage. Infection prevention and control (IPC), including the use of personal protection equipment (PPE), and measures for patient transport will follow national guidelines in each country. Written informed consent/assent will be sought. The study is anticipated to start in January 2021 and last for approximately 18 months.

DETAILED DESCRIPTION:
Background: In Africa, COVID-19 has the potential to cripple the continent's fragile healthcare systems and be devastating economically. It is unknown whether malaria infection worsens COVID-19, affects the acquisition of protective antibodies against the SARS-CoV-2 virus, or contributes to its onwards spread by resulting in higher viral loads and/or longer duration of viral shedding. It is also unknown if the effective clearance of malaria parasites and/or the choice of antimalarials affects any of these potential associations. His study will determine if the antimalarial pyronaridine, in the fixed-dose combination of pyronaridine-artesunate, has a positive, negative or negligible effect on COVID-19 disease progression or duration of viral carriage and the seroconversion rate to SARS-CoV-2.

Methods: A malaria treatment trial will be conducted nested within a larger observational COVID-19 cohort study in highly malaria-endemic areas in western Kenya and Burkina-Faso. The COVID-19 cohort study consists of approximately 708 newly diagnosed COVID-19 patient of all ages. They will be enrolled from a source population of approximately 4,720 individuals of all ages screened for SARS-CoV-2. It is anticipated that approximately 142 of the 708 cohort participants will be co-infected with malaria. These co-infected participants will be enrolled in the nested malaria treatment trial if they have uncomplicated malaria and are able to take oral medication. They will be randomized to receive either a standard 3-day treatment course of artemether-lumefantrine (the current first-line treatment) or pyronaridine-artesunate, a new highly effective antimalarial combination that is being rolled out as first or second-line treatment in western Kenya and Burkina Faso. All 142 patients will be followed for 42 days and nasal swabs and blood samples taken on days 1, 3, 7, 14, and 28. Malaria smears will be taken on days 3, 7, 14, 21, 28 and 42. The primary endpoint is the rate of SARS-CoV-2 clearance by day-7.

To limit the transmission of SARS-CoV-2, strict adherence to infection prevention and control (IPC) guidelines, including use of personal protection equipment (PPE), and measures for patient transport will be followed as per national guidelines in each country. Written informed consent/assent will be sought.

Partners: This 18-months study is funded by the Bill and Melinda Gates Foundation and is part of a collaboration between the Kenyan Medical Research Institute (KEMRI) in Kenya; the US Centers for Disease Control and Prevention (CDC); the Liverpool School of Tropical Medicine (LSTM); the Ministry of Health, Kenya; the Groupe de Recherche Action en Santé (GRAS), Ouagadougou, Burkina Faso; the Ministry of Health in Burkina Faso, and the London School of Hygiene and Tropical Medicine (LSHTM). LSTM and LSHTM will act as sponsors for the studies in Kenya and Burkina Faso, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmed SARS-CoV-2 infection, with positive molecular test results within the past 72 hours*
* Aged >=6 months **
* Resident in the study area
* The participant or caretaker is willing and able to give informed consent or assent with parent/guardian informed consent for participation in the study
* Agrees not to self-medicate with chloroquine, hydroxychloroquine or other antimalarials with potential anti-SARS-CoV-2 properties
* Not previously diagnosed with COVID-19
* Contactable by phone for follow-up permitting real-time, reliable information
* Uncomplicated malaria, defined as able to take oral medication
* Bodyweight ≥5kg
* Confirmed malaria infection by RDT (pLDH) or microscopy

Exclusion Criteria:

* Unwilling or unable to provide informed consent/assent
* The participant is judged by the Investigator to be at significant risk of failing to comply with the provisions of the protocol as to cause harm to self or seriously interfere with the validity of the study results
* Inability/unlikely to be in the study area for the duration of the 28-day follow-up period
* Pregnant or lactating women
* Severe disease requiring parenteral treatment
* Currently receiving, or recently received (within the last 28 days) pyronaridine-artesunate or artemether-lumefantrine
* Received chloroquine in the last three days
* Inability/unlikely to be in the study area for the duration of the 42-day follow-up period
* Known hypersensitivity or specific contraindication to the use of any of the study drugs in the treatment arms
* Known chronic kidney disease (signs or symptoms of stage IV renal impairment or receiving dialysis)
* Known liver cirrhosis (Child-Pugh Class B or greater) or signs or symptoms of severe hepatotoxicity

Ages: 6 Months to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Incidence of SARS-CoV-2 clearance | by day 7
  Defined as the proportion of participants with a negative nasal swab on Day 7 after the start of treatment

SECONDARY OUTCOMES:
Median viral load of SARS-CoV-2 | by day 14
  Median CT value as detected from mid-nasal swabs by PCR
Cumulative incidence of SARS-CoV-2 clearance | by days 14, 21 and 28
  Defined as the proportion of participants with negative nasal swabs
Time to clearance of nasal SARS-CoV-2 | by days 1, 3, 7, 14 and 28
  Defined as the number of days to a negative SARS-CoV-2 RNA PCR tests (swabs collected on days 1, 3, 7, 14, 21 and 28)
Cumulative seroconversion rates (IgG, IgM, IgA) | by days 7, 14, 21 and 28
  proportion of antibody negative patients on enrolment who seroconvert
IgG, IgM, IgA antibody titres against SARS-CoV-2 | by days 7, 14, 21 and 28
  Geometric mean, maximum, and change from baseline
IL-6, IL-7, IL-10, TNF-alpha and Interferon-Gamma | by days 3, 7, 14 and 28
  median, max and change from baseline
CRP and angiotensin-2, angiopoietin-1 and angiopoietin-2 | by days 3, 7, 14 and 28
  median, max and change from baseline
Genomic responses to SARS-CoV-2 infection | by day 28
  Transcriptional profiling (gene expression) of whole blood and fixed whole blood for T and B cell markers
Cellular immune responses to SARS-CoV-2 infection | by day 28
  T cell responses
The clinical and parasitological antimalarial treatment response | by day 42
  Expressed as the proportion with early treatment failure, late clinical failure, late parasitological failure or an adequate clinical and parasitological response. Recrudescence will be differentiated from new infection by genotyping of malaria parasites
COVID-19 disease severity | by day 28
  Defined by a severity index score for COVID-19
COVID-19 disease duration | by day 28
  The proportion of days with symptoms after randomization
COVID-19 fever duration | by day 28
  The proportion of days with a fever after randomization
COVID-19 respiratory symptoms duration | by day 28
  The proportion of days with respiratory symptoms after randomization
COVID-19 disease duration in days | by day 28
  The number of days until symptom clearance
Treatment-related adverse events, serious adverse events, and adverse events resulting in treatment discontinuation | by day 7
  The cumulative proportion of patients with any of these events after the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kariuki Simon, PhD, Principal Investigator — Kenya Medical Research Institute; Sirima Sodiomon, MD, PhD, Principal Investigator — Groupe de Recherche Action en Sante
Locations (2):
- Ouagadougou Hospitals, Ouagadougou, Burkina Faso
- Kisumu County Referral Hospital, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
We will encourage data sharing to ensure that the scientific potential of this study is maximized. The full anonymized research database will be made publicly available as soon as the full study findings have been published or based on any data requests that may occur during the study or analysis is still ongoing. For the databases, we will use a controlled access approach.
Supporting Information: Study Protocol
Time Frame: As soon as the full study findings have been published or based on any data requests that may occur during the study or analysis is still ongoing.
Access Criteria: Data access will be provided to researchers after a proposal has been approved by an independent review committee identified for this purpose. An agreement on how to collaborate will be reached based on any overlap between the proposal and any ongoing efforts. Proposals can be directed to email addresses provided in the publications and websites. To gain access, data requesters will need to sign a data-sharing agreement. The only limits to data sharing will be to safeguard research participants' confidentiality. External users will be bound by data-sharing agreements in line with the Data Sharing Policy from the respective Sponsors and the Gates Foundation to ensure that the privacy of individuals is protected. The agreement will prohibit any attempt to (a) identify study participants from the data or otherwise breach confidentiality, (b) make unapproved contact with study participants.

REFERENCES:
- [Derived] Tangara B, Barsosio HC, Marlais T, Kabore JMT, Tiono AB, Otieno K, Wanjiku M, Achieng M, Onyango ED, Ondieki ED, Aura H, Odawo T, Allen DJ, Hannan L, Tetteh KK, Soulama I, Ouedraogo A, Serme SS, Soulama BI, Barry A, Badoum ES, Matthewman J, Brazal-Monzo H, Canizales J, Drabko A, Wu W, Kariuki S, Lesosky M, Sirima SB, Drakeley C, Ter Kuile FO. Artemether-lumefantrine versus pyronaridine-artesunate for the treatment of malaria in patients with mild to moderate COVID-19 in Kenya and Burkina Faso: a randomised open-label trial (MALCOV). EClinicalMedicine. 2026 Jan 3;91:103735. doi: 10.1016/j.eclinm.2025.103735. eCollection 2026 Jan. PMID 41552003